CLINICAL TRIAL: NCT01764984
Title: Randomized Clinical Evaluation of Bone Mineral Density Changes Under Non-cemented Trabecular Metal Tibial Component and Cemented Titanium Controls.
Brief Title: Bone Mineral Density Changes Under Two Tibial Components in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Étienne Belzile, Principal Investigator; Orthopaedic surgeon, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5.5.04.12
Record Dates: First submitted 2012-02-17; First posted 2013-01-10 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Unilateral Primary Osteoarthritis of Knee
Keywords: total knee arthroplasty; trabecular metal; bone mineral density
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabecular metal (Experimental): Primary Total Knee Arthroplasty is performed with a non cemented trabecular metal tibial baseplate.
  Interventions: Device: Total knee arthroplasty
- Titanium (Active Comparator): Primary total knee arthroplasty is performed with cemented titanium traditional tibial base plate
  Interventions: Device: Total knee arthroplasty

INTERVENTIONS:
Device: Total knee arthroplasty — Total knee arthroplasty using parapatellar approach and postero-stabilized implants.
  Other Names: NexGen LPS Monobloc (Trabecular Metal) tibia (Zimmer); NexGen Option Stemmed (Titanium) modular tibia (Zimmer).

SUMMARY:
Osteoarthritis is a progressive disease afflicting to two thirds of Americans. Today, an estimated 43 million individuals have arthritis. By 2020, more than 59.4 million Americans will be affected by the disease. Despite the relative good track record of total knee replacement, it remains a biomedical device that can fail over time. A recent study looking at the current mechanisms of total knee replacement failures, listed polyethylene wear and osteolysis around implants. The material used for polyethylene insert as well as the conformity of articular surface of implants has been modified to decrease wear. While introducing modularity, the usage of metal backing in tibial base plates became obvious as it offered better stress distribution to the proximal tibial bone. However, it introduced other modes of failures. Micromotion has been demonstrated between the metal backing and the tibial liner, and produced backside polyethylene wear in 44% of implants at retrieval for revision. Factor influencing the surgeon's choice of implant include: reproductibility and longevity of results, technical difficulty of implantation, cost, and impact on bone stock. The modulus of elasticity of the tibial base plate has a direct effect on periprosthetic bone biology. Studies have described a significant decrease in postoperative Bone mineral density (BMD), adjacent to the implants, after total knee replacement. No study, to our knowledge, has looked at BMD in vivo after total knee replacement comparing different tibial base plate designs. Direct effect of changes in design on overall implant survival can be studied with randomized clinical trials isolating specific variables. No randomized clinical trial has looked at tibial insert stiffness and modularity, and it effect on bone density changes, synovitis, osteolysis or survivorship. In order to isolate stiffness and modularity as study variables, one would aim at randomizing an homogenous patient population undergoing total knee arthroplasty with implants of similar articular geometry designs with different tibial insert modularity and stiffness.

DETAILED DESCRIPTION:
Number of patients: 80 Ages: 55 - 75 years old Sex: male and female Race: all

ELIGIBILITY:
Inclusion Criteria:

* Tri-compartmental knee arthrosis
* 55 to 75 years of age
* Stable health condition

Exclusion Criteria:

* Inflammatory arthritis
* Osteonecrosis
* Infection
* Amputation (AK or BK)
* Biphosphonates
* Metal in the proximal tibia (25cm)
* History of fracture or osteotomy
* Ligament instability

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-11; Primary Completion 2009-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mineral Density (%) from baseline initial value | post-operative 7 to 10 days, 6,12,24 months
  Evaluation of Bone Mineral Density using dual energy x-ray absorptiometry (DEXA) scan under tibial base plate implant after Total knee arthroplasty.

SECONDARY OUTCOMES:
Western Ontario & McMAster University Osteoarthritis sCore (WOMAC)change in time. | Pre-operative, 6,12,24,60 months
  Standardized clinical evaluation instrument specific to Total knee arthroplasty population.
number of study subject with implant loosening | 12, 24, 60 months
  Radiological evaluation of implant loosening according to Radiographic Knee Society Score at follow-up after total knee arthroplasty.
Knee injury and Osteoarthritis Outcome Score (KOOS) change in time. | pre-operative, 6,12,24,60 months
  Standardized clinical outcome instruments specific to total knee arthroplasty population.
SF-36 score | Pre-operative, 12,24,60 months
  Standardized General health evaluation and quality of life measuring instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne L Belzile, MD, Principal Investigator — Centre Hospitalier Universitaire de Quebec - Universite Laval
Locations (3):
- Canada (3):
  - Hôpital Maisonneuve Rosemont, Montreal, Quebec
  - Hopital du Sacre-Coeur, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec